CLINICAL TRIAL: NCT01138813
Title: Development of Magnetic Resonance Spectroscopy (MRS) Biomarkers of Tumor Metabolism
Brief Title: Development of Magnetic Resonance Spectroscopy (MRS) Biomarkers of Tumor Metabolism (MK-0000-145)
Acronym: MRS Tumor
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0000-145; 145; 2010_027
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Glioma
Keywords: magnetic resonance spectroscopy (MRS); lactate editing; metabolite content; glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Male and female patients aged 18-70 years old with newly diagnosed operable glioma of grade II or higher

SUMMARY:
This study will evaluate the test-retest repeatability of lactate and other metabolites measured by single voxel magnetic resonance spectroscopy (MRS) and multi-voxel magnetic resonance spectroscopic imaging experiments (MRSI) in tumor tissue in patients radiographically diagnosed with glioma.

These measurements will test whether the concentration of lactate in tumor will be higher than the concentration of lactate in normal tissue of the same patient.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18-70 years old with newly diagnosed operable glioma of grade II or higher which is > 3cm in diameter based on radiographic examination
* Patients about to receive biopsy or resection of newly diagnosed glioma

Exclusion Criteria:

* Contraindication to magnetic resonance imaging (MRI): e.g. cardiac pacemaker, metallic implants, known contrast allergy, and pregnancy
* Impaired renal function
* Current or previous chemotherapy, radiation, or other tumor treatment excluding steroids
* Tumor location extra-cerebral, temporal, or in close proximity to frontal sinus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients aged 18-70 years old with newly diagnosed operable glioma of grade II or higher
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The test-retest repeatability of lactate and other metabolites when measured by multi-voxel MRSI in tumor tissue | 90 minutes
The test-retest repeatability of lactate and other metabolites when measured by single voxel MRS | 90 minutes

SECONDARY OUTCOMES:
The geometric mean fold rise (GMFR) in the concentrations of lactate and each of the other metabolites for tumor/normal tissue | 90 minutes
The test-retest repeatability of lactate and other metabolites when measured by multi-voxel MRSI in normal tissue | 90 minutes
True geometric mean ratio (GMR) of the MRSI/SV MRS concentration values | 90 minutes
The mean levels of each of the metabolites will be summarized by tumor grade and type | 90 minutes
The correlation between in vivo (measured by MRSI) and in vitro levels of lactate and other metabolites in tumors | 90 minutes
The within day and between day standard deviations for each metabolite | 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] McLean MA, Sun A, Bradstreet TE, Schaeffer AK, Liu H, Iannone R, Herman G, Railkar RA, Joubert I, Gillard JH, Price SJ, Griffiths JR. Repeatability of edited lactate and other metabolites in astrocytoma at 3T. J Magn Reson Imaging. 2012 Aug;36(2):468-75. doi: 10.1002/jmri.23673. Epub 2012 Apr 25. PMID 22535478